CLINICAL TRIAL: NCT03435055
Title: Network-Level Effects of Nitrous Oxide in the Human Brain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Richard Harris, Associate Professor of Anesthesiology and Associate Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00096321
Record Dates: First submitted 2018-01-25; First posted 2018-02-15 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — Endothelium-Dependent Relaxing Factors; Inhalation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nitrous Oxide - inhaled (Experimental): Each volunteer will participate in one scanning visit in which simultaneous functional magnetic resonance imaging (fMRI) and electroencephalogram (EEG) data will be collected wherein they receive placebo (20 minutes) followed by inhaled nitrous oxide at subanalgesic levels (35% inhaled concentration) over 40 minutes.
  Interventions: Drug: Nitrous Oxide Gas for Inhalation

INTERVENTIONS:
Drug: Nitrous Oxide Gas for Inhalation — Each volunteer will participate in one scanning visit in which simultaneous functional magnetic resonance imaging (fMRI) and electroencephalogram (EEG) data will be collected wherein they receive placebo (20 minutes) followed by inhaled nitrous oxide at subanesthetic levels (35% inhaled concentration) over 40 minutes.

SUMMARY:
The purpose of this study is to understand how a commonly used drug, nitrous oxide, acts on the brain to reduce pain. Nitrous oxide is commonly used in anesthesiology but there is limited knowledge on how this drug affects functional networks in the brain.

DETAILED DESCRIPTION:
The objective of this study is to identify the network transformations that account for the analgesic effects of nitrous oxide. Our hypothesis is that analgesic doses of nitrous oxide increase network efficiency and disrupt normal pain processingOur approach is to administer subanesthetic nitrous oxide during the acquisition of fMRI (functional magnetic resonance imaging) and EEG (electroencephalogram).

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index <30
2. Must be right-handed
3. Must be capable of giving written informed consent

Exclusion Criteria:

1. History of obstructive sleep apnea;
2. History of a difficult airway with a previous anesthetic
3. Gastroesophageal reflux;
4. Hypertension or other cardiovascular abnormalities;
5. Pulmonary hypertension;
6. History of recreational drug use;
7. History of chronic alcohol abuse
8. Having any chronic medical illness involving pain;
9. History of major depression;
10. History of psychosis or bipolar disorder;
11. History of methylenetetrahydrofolate reductase deficiency;
12. History of a known hypersensitivity to ketamine, midazolam, Zofran, labetalol or glycopyrrolate
13. History of seizures or other neurologic disorders;
14. Pregnant or nursing mothers;
15. Tattoos on the head or neck region - all other tattoos are subject to determination by investigators;
16. Contraindications to neuroimaging methods;
17. Any impairment, activity or situation that in the judgment of the Study Coordinator or Principal Investigators would prevent satisfactory completion of the study protocol.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Harris, PhD, Principal Investigator — Associate Professor of Anesthesiology and Associate Professor of Internal Medicine
Locations (1):
- Michigan Medicine - University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dai R, Larkin TE, Huang Z, Tarnal V, Picton P, Vlisides PE, Janke E, McKinney A, Hudetz AG, Harris RE, Mashour GA. Classical and non-classical psychedelic drugs induce common network changes in human cortex. Neuroimage. 2023 Jun;273:120097. doi: 10.1016/j.neuroimage.2023.120097. Epub 2023 Apr 7. PMID 37031827

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 21 participants consented to participate but 2 participants did not participate in any part of the research.
Groups:
- Nitrous Oxide - Inhaled: Each volunteer will participate in one scanning visit in which simultaneous fMRI/EEG data will be collected wherein they receive placebo (20 minutes) followed by inhaled nitrous oxide at subanalgesic levels (35% inhaled concentration) over 30 minutes.
Period: Screening
Arm/Group | Nitrous Oxide - Inhaled
Started | 21
Completed | 19
Not Completed | 2
Not completed — Physician Decision | 2
Period: Received Intervention
Arm/Group | Nitrous Oxide - Inhaled
Started | 19
Completed | 16
Not Completed | 3
Not completed — Did not complete nitrous administration | 3

BASELINE CHARACTERISTICS:
Arm/Group | Nitrous Oxide - Inhaled
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] — Average age of participant, continuous
  years | 25 [20 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Functional Connectivity During Nitrous Oxide
Description: Functional connectivity measures will be assessed at rest (baseline) and during sub anesthetic dose nitrous oxide (nitrous oxide). Seed-to-whole brain functional connectivity (Fisher's r-transformed z) will be measured from the left anterior insula, previously shown to be involved in pain and sensory processing. Paired t-test were conducted on subject specific beta maps to identify changes in connectivity associated with nitrous oxide in SPM12. The z-score descriptors represent the Fishers-r-to-z transformed. Here the z-score is a transformation of the Pearson's (r) correlation coefficient of the BOLD timeseries between two brain regions. Higher z-scores are associated with higher correlations in timeseries and correspond with higher functional connectivity between two brain regions.
Time Frame: Baseline to 50 minutes
Population: Three participants had missing data because they did not complete the full scanning protocol.
Measure: Mean (Standard Deviation); unit: Fisher's r transformed z score
Groups:
- Pre-Nitrous: Each volunteer will participate in one scanning visit in which simultaneous fMRI/EEG data will be collected as they receive oxygen (20 minutes) followed
  Functional connectivity (Fisher's r to z transformed) between the left anterior insula and superior frontal gyrus were measured at baseline.
- Nitrous Oxide - Subanesthetic Dose: Each volunteer will participate in one scanning visit in which simultaneous fMRI/EEG data will be collected as they received subanesthetic dose of nitrous oxide at (35% inhaled concentration) over 30 minutes.
  Functional connectivity (z-score) between the left anterior insula and superior frontal gyrus were measured during administration of subanesthetic nitrous oxide.
Arm/Group | Pre-Nitrous | Nitrous Oxide - Subanesthetic Dose
Number analyzed (Participants) | 16 | 16
Fisher's r transformed z score
  L superior frontal gyrus | 0.1123 (0.0639) | 0.0358 (0.0620)
  R superior frontal gyrus | 0.1492 (0.1179) | 0.0394 (0.0950)
Statistical Analysis 1: Comparison: Pre-Nitrous vs Nitrous Oxide - Subanesthetic Dose; Paired t-test were conducted on subject specific beta maps to identify changes in connectivity associated with nitrous oxide in SPM12. Hypothesis was that the results would be deemed significant at false discovery rate (FDR) cluster level corrected p < 0.05 derived from a voxel-wise uncorrected p-value < 0.001; Test type: Superiority; p = 0.001, t-test, 2 sided

2. Primary Outcome: Functional Connectivity Associated With Tonic Stimulus
Description: Functional connectivity measures will be assessed at rest (baseline) and during a tonic cuff stimulus (6-minutes). Seed-to-whole brain functional connectivity (Fisher's r-transformed z) will be measured from the left anterior insula, previously shown to be involved in pain and sensory processing. Paired t-test were conducted on subject specific beta maps to identify changes in connectivity associated with nitrous oxide in SPM12. The z-score descriptors represent the Fishers-r-to-z transformed. Here the z-score is a transformation of the Pearson's (r) correlation coefficient of the BOLD timeseries between two brain regions. Higher z-scores are associated with higher correlations in timeseries and correspond with higher functional connectivity between two brain regions.
Time Frame: Baseline to 50 minutes
Population: Number of participants scanned.
Measure: Mean (Standard Deviation); unit: Z score
Groups:
- Pre-Tonic Cuff: Each volunteer will participate in one scanning visit in which simultaneous fMRI/EEG data will be collected as they receive oxygen (20 minutes) at rest and during a tonic cuff stimulus applied to the leg (6 minutes).
  Functional connectivity (Fisher's r to z score transformed) between the left anterior insula and the postcentral gyrus prior to (baseline) and during a tonic cuff stimulus.
- Tonic Cuff Stimulus: Each volunteer will participate in one scanning visit in which simultaneous fMRI/EEG data will be collected while a tonic cuff stimulus was applied to the calf of the left leg (6 minutes).
  Functional connectivity (z score) was measured between the left anterior insula and the right postcentral gyrus from the fMRI data during the tonic cuff stimulus.
Arm/Group | Pre-Tonic Cuff | Tonic Cuff Stimulus
Number analyzed (Participants) | 19 | 19
Z score | -0.0509 (0.0822) | 0.0486 (0.1001)
Statistical Analysis 1: Comparison: Pre-Tonic Cuff vs Tonic Cuff Stimulus; Paired t-test were conducted on subject specific beta maps to identify changes in connectivity associated with nitrous oxide in SPM12. Hypothesis was that results would be deemed significant at false discovery rate (FDR) cluster level corrected p < 0.05 derived from a voxel-wise uncorrected p-value < 0.001; Test type: Superiority; p = 0.006, t-test, 2 sided

3. Secondary Outcome: Tonic Stimulus Intensity During Nitrous Oxide
Description: Participants will receive a tonic (6 minutes) pressure applied to the lower leg at baseline and under subanesthetic dose of nitrous oxide (35% inhaled concentration). Following each pressure stimulus, participants will rate the pain intensity of the tonic stimulus (0 ="no pain", 10= "worst pain imaginable", Visual Analog Scale, e.g pain intensity).
Time Frame: Baseline to 50 minutes
Population: Three participants had missing data because they did not complete the full scanning protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-nitrous; Nitrous Oxide - 35% Inhaled Concentration: Participants will receive a tonic (6 minutes) pressure applied to the lower leg prior to (baseline) and during administration of subanesthetic dose of nitrous oxide (35% inhaled concentration). Following each pressure stimulus, participants will rate the pain intensity of the tonic stimulus (0 = "no pain", 10= "worst pain imaginable", Visual Analog Scale, e.g pain intensity.
Arm/Group | Pre-nitrous | Nitrous Oxide - 35% Inhaled Concentration
Number analyzed (Participants) | 16 | 16
score on a scale | 4.9688 (1.217) | 2.500 (2.309)
Statistical Analysis 1: Comparison: Pre-nitrous vs Nitrous Oxide - 35% Inhaled Concentration; Paired-t tests were conducted to determine whether changes in stimulus intensity: post stimulus at baseline and under subanesthetic dose of nitrous oxide. Statistical tests were completed in SPSS 26 and determined by p < 0.05; Test type: Superiority; p < 0.01, t-test, 2 sided

4. Secondary Outcome: Spectral Power of Sub-anesthetic Dose of Nitrous Oxide
Description: Brain imaging data were obtained from functional magnetic resonance imaging (fMRI) data recorded simultaneously with electroencephalography (EEG) data at baseline and under a sub-anesthetic dose of nitrous oxide. Spectral data were averaged from EEG data at all electrodes collected during the baseline and sub-anesthetic dose (35%) of nitrous oxide to observe changes in spectral power. The EEG power spectrum was divided into three frequency bands: Delta = 1-3 Hz; Theta = 4-7 Hz; and Alpha = 8 - 13 Hz
Time Frame: Baseline to 50 minutes
Measure: Mean (Standard Deviation); unit: dB (decibels)
Groups:
- Pre-Nitrous: Each volunteer will participate in one scanning visit in which simultaneous fMRI/EEG data will be collected as they receive oxygen (20 minutes) followed
- Nitrous Oxide - Subanesthetic Dose: Each volunteer will participate in one scanning visit in which simultaneous fMRI/EEG data will be collected as they received subanesthetic dose of nitrous oxide at (35% inhaled concentration) over 30 minutes.
Arm/Group | Pre-Nitrous | Nitrous Oxide - Subanesthetic Dose
Number analyzed (Participants) | 16 | 16
dB (decibels)
  Delta | 13.31 (2.20) | 14.65 (2.56)
  Theta | 11.88 (1.89) | 12.80 (1.87)
  Alpha | 6.72 (1.92) | 6.97 (2.05)
Statistical Analysis 1: Comparison: Pre-Nitrous vs Nitrous Oxide - Subanesthetic Dose; Delta; Test type: Other — Paired T-test comparing baseline to nitrous; p = 0.0622, Paired t-test
Statistical Analysis 2: Comparison: Pre-Nitrous vs Nitrous Oxide - Subanesthetic Dose; Theta; Test type: Other — Paired T-test comparing baseline to nitrous; p = 0.0292, Paired t-test
Statistical Analysis 3: Comparison: Pre-Nitrous vs Nitrous Oxide - Subanesthetic Dose; Alpha comparison; Test type: Other — Paired T-test comparing baseline to nitrous; p = 0.5905, Paired t-test

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 24 hours.
Description: The definition of adverse event and/or serious adverse event does not differ from the clinicaltrials.gov definition.
Groups:
- Nitrous Oxide - Inhaled: Each volunteer will participate in one scanning visit in which simultaneous fMRI/EEG data will be collected wherein they receive placebo (20 minutes) followed by inhaled nitrous oxide at subanalgesic levels (35% inhaled concentration) over 30 minutes.
  A total of 21 participants consented to participate but 2 participants did not participate in any part of the research and thus no adverse events data could have been collected.
Arm/Group | Nitrous Oxide - Inhaled
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 2/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrous Oxide - Inhaled (N=19)
Tachycardia (General disorders) | 1 (1) — Tachycardia
Emesis (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Data for the Spectral Power of Sub-anesthetic Dose of Nitrous Oxide outcome measure will be analyzed within the coming year and the ClinicalTrials.gov record will be updated at that time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT03435055/Prot_SAP_000.pdf